CLINICAL TRIAL: NCT00724529
Title: Post Marketing Surveillance of Remicade in Inflammatory Bowel Disease (IBD)
Brief Title: Post Marketing Surveillance of Remicade
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100771; REMICADECRD4015 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Crohn's Disease; Ankylosing Spondylitis
Keywords: Crohn's Disease; Ankylosing Spondylitis
MeSH Terms: conditions — Crohn Disease; Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Serious Active Crohns Disease: Patients with severe active Crohns Disease who do not show any response to treatment with corticosteroids or immunosuppressive agents, and have no drug tolerance or contraindications to such treatments.
  Interventions: Biological: Infliximab
- Fistula-Type Active Crohns Disease: Patients with fistula-type Crohns Disease who do not show any response to general treatments such as antibiotics, drainage, or immunosuppressant.
  Interventions: Biological: Infliximab
- Ankylosing Spondylitis: Patients with Ankylosing Spondylitis who do not show adequate response to general treatments and with increased serological indices related to severe axial symptoms and inflammation.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg IV given in a schedule according to the official label, based on the indication it is being used for.
  Other Names: SCH 215596; Remicade

SUMMARY:
The purpose of this study is to understand the safety and effectiveness of infliximab when used in clinical practice. This is a post-marketing surveillance study.

DETAILED DESCRIPTION:
The investigator will record continuously from the first patient since the day of contract to the numbers of patients of contract based on Remicade approval.

ELIGIBILITY:
Inclusion Criteria:

* Severe active Crohn's disease: the patients with severe active Crohn's disease who do not show any response to the treatment with corticosteroid or immunosuppressive agents, have no drug tolerance, or are contraindicated to such treatments.
* Fistula-type active Crohn's disease: the patients with fistula-type active Crohn's disease who do not show any response to general treatments such as antibiotics, drainage, or immunosuppressant.
* Ankylosing spondylitis: the patients with ankylosing spondylitis who do not show adequate response to general treatments, and with increased serological indices related to severe axial symptoms and inflammation.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of subjects will mainly be taken from the digestive or rheumatoid departments of internal medicine in university or general hospitals, where patients with Crohn's Disease and Ankylosing Spondylitis are generally treated. The period of surveillance is from 23 AUG 2005 to 22 AUG 2011.
Sampling Method: Probability Sample
Enrollment: 938 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of Remicade Injection (Infliximab) when used in clinical practice | The maximum period for observation in this surveillance would be 30 weeks (6 administrations) for patients with Crohn's disease and 24~30 weeks (6 administrations) for patients with Ankylosing spondylitis.

SECONDARY OUTCOMES:
To evaluate the efficacy of Remicade Injection (Infliximab) when used in clinical practice | The maximum period for observation in this surveillance would be 30 weeks (6 administrations) for patients with Crohn's disease and 24~30 weeks (6 administrations) for patients with Ankylosing spondylitis.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea